CLINICAL TRIAL: NCT01170234
Title: Exhaled Nitric Oxide as a Biomarker of Disease Activity in Eosinophilic Esophagitis
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: TUFTS-EOE-FENO
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Eosinophilic Esophagitis
Keywords: Exhaled nitric oxide; Eosinophilic esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eosinophilic esophagitis (EoE): Treatment-naïve EoE patients, age 7 -65
  Interventions: Device: NIOX MINO® Airway Inflammation Monitor

INTERVENTIONS:
Device: NIOX MINO® Airway Inflammation Monitor — We will measure exhaled nitric oxide of patients with eosinophilic esophagitis pre-, during and post- treatment at pre-defined time intervals.

SUMMARY:
There is currently no reliable, noninvasive biomarker for eosinophilic esophagitis (EoE), a chronic allergic diseases characterized by significant infiltration of eosinophils in the esophagus. Because eosinophils release nitric oxide, levels of exhaled nitric oxide (FeNO) are used routinely for guiding treatment in subsets of patients with asthma. FeNO levels are also elevated in immunological diseases that do not involve the airways. The investigators hypothesize that patients with EoE have elevated nitric oxide concentration in their exhaled breath and that changes in FeNO levels could be used to measure disease activity. The objective of this study is to determine the feasibility of using FeNO as a noninvasive surrogate marker for EoE disease activity. The investigators propose to measure serial exhaled nitric oxide (FeNO) levels on a group of patients with confirmed EoE, before, during and after the course of topical corticosteroid therapy to determine whether the level declines from pre-treatment level in individual patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-65.
* Confirmed diagnosis of EoE. The diagnosis of eosinophilic esophagitis is based upon the presence of characteristic clinical features and large numbers of eosinophils in the esophagus on pathologic examination (≥15 eosinophils per high powered [400x] field in at least one specimen) despite acid suppression with a PPI for one to two months. The criteria also include normal gastric and duodenal mucosal biopsies and the exclusion of other causes. Clinical features in adults include dysphagia, pain and/or history of food impaction. Symptoms in children vary depending in part upon their age: feeding disorders (median age 2.0), vomiting (median age 8.1), abdominal pain (median age 12.0), dysphagia (median age 13.4), and food impaction (median age 16.8).

Exclusion Criteria:

* Use of systemic or inhaled corticosteroids in the preceding 3 months.
* History of doctor-diagnosed asthma, acute or chronic rhinosinusitis.
* History of cirrhosis.
* History of kidney, heart or lung disease.
* Pregnancy

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gastroenterology outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Exhaled nitric oxide as a biomarker for disease activity in eosinophilic esophagitis | 2 years
  The objective of this study is to determine the feasibility of using exhaled nitric oxide (FeNO) as a noninvasive surrogate marker for EoE disease activity. We will measure FeNO levels on a group of patients with confirmed EoE before, during and after the course of topical corticosteroid therapy.
Exhaled nitric oxide as a biomarker for disease activity in eosinophilic esophagitis | 2 years
  Change in exhaled nitric oxide levels during corticosteroid treatment.

SECONDARY OUTCOMES:
Exhaled nitric oxide as a biomarker for disease activity in eosinophilic esophagitis | 2 years
  Intra- and inter-patient variability in exhaled nitric oxide levels.

CONTACTS AND LOCATIONS:
Overall Officials: John Leung, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Recommendations for standardized procedures for the on-line and off-line measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide in adults and children-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 1999 Dec;160(6):2104-17. doi: 10.1164/ajrccm.160.6.ats8-99. No abstract available. PMID 10588636